CLINICAL TRIAL: NCT06144307
Title: Effects of External Oblique Fascial Plan Block and Subcostal Transversus Abdominis Plan Block on Postoperative Pulmonary Functions
Brief Title: Effects of Fascial Plan Blocks on Pulmonary Functions
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Bengü Gülhan Köksal, Principal Investigator, Zonguldak Bulent Ecevit University
Other Study IDs: 2023/04-3
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Pain, Postoperative; Respiratory Function Loss
Keywords: postoperative pain; plane block; pulmonary function
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- External Oblique Fascial Plan Block
  Interventions: Procedure: plane block
- Subcostal Transversus Abdominis Plan Block
  Interventions: Procedure: plane block
- Control

INTERVENTIONS:
Procedure: plane block — injection of local anesthetic to the myofascial plane
  Groups: External Oblique Fascial Plan Block; Subcostal Transversus Abdominis Plan Block

SUMMARY:
In addition to the traumatic effect of the operation, the effort to immobilize the auxiliary respiratory muscles due to pain causes a decrease in postoperative respiratory function (especially in thoracic and upper abdominal surgeries). In addition, superficial and tachypneic breathing caused by the inability of the patient to take deep breaths with pain leads to closure of small airways and increase in intrapulmonary shunts, resulting in hypoxia. Postoperative pain management is important not only to prevent pain but also to reduce pulmonary complications that may occur due to changes in lung function and to reduce mortality and morbidity by controlling the stress response. Pain after nausea and vomiting is the most common reason for hospitalization after laparoscopic surgery.

Although pain in laparoscopic cholecystectomy (LC) has many components including incisional, visceral and reflected, the primary source of pain is incisional pain. A multimodal analgesic approach (NSAII, paracetamol, opioids, local infiltration, facial plane blocks and paravertebral and periparavertebral blocks) is recommended. Regional anesthesia combined with general anesthesia reduces the stress response associated with surgery and reduces the need for opioid use. Subcostal TAP Block; injection of local anesthetic between the internal oblique and transversus abdominis muscles in the upper quadrant of the anterior abdominal wall blocks the anterior cutaneous branches of the thoracoabdominal nerves. External Oblique Fascial Plane Block (EOIB); blocks both the anterior and lateral cutaneous branches of the thoracoabdominal nerves. It is performed between the 6th-7th costae. There is a cutaneous sensory block between T6-T9 in the midabdomen and T6-T10 in the anterior axillary line.

The conventional method is the administration of intravenous opioids as a method of postoperative analgesia when the routine block cannot be performed due to a contraindication.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* ASA I-II-III risk group
* Patients whose consent was obtained with an informed consent form
* She will undergo a cholecystectomy operation
* Patients to be cooperative for SFT test

Exclusion Criteria:

* <18 years and >65 years
* ASA ≥ IV
* Pulmonary function test below 50% of the expected value
* Known diaphragm paralysis
* Body mass index >30
* Myocardial infarction within 1 month
* Dementia or confusion
* Lack of cooperation
* People with respiratory diseases
* Congestive heart failure
* Unstable hypertension
* Thoracoabdominal surgery

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo cholecystectomy between the ages of 18-65
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
the effect of plane blocks on postoperative pulmonary function | during the postoperative 24 hours
  The effect of pain relief after plane blocks on postoperative pulmonary function

SECONDARY OUTCOMES:
opioid consumption | during the postoperative 24 hours
  need for opioids as a result of pain
Incidence of nausea and vomiting | during the postoperative 24 hours
  Need for nausea and vomiting
quality of recovery-15 | during the postoperative 24 hours
  Quality of recovery of patients by survey

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Faculty of Medicine, Kozlu, Zonguldak Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No